CLINICAL TRIAL: NCT06943222
Title: Comparative Effects of Traditional Play and Free Play on Motor Fitness and Social Interaction in Primary School Children
Brief Title: Comparative Effects of Traditional Play and Free Play in Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/0741
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Children
Keywords: Childhood; Motor skills; Social skills; Traditional games
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Play (Experimental): Traditional play groups will partake in organized conventional activities that are included in their schedule
  Interventions: Other: Traditional Play
- Free play (No Intervention): free play groups will involve themselves in unregulated spontaneous play. The participants will be segregated into 2 distinct groups. The flamingo balance tests (FLA) will be used to assess motor fitness related to balance; the standing long jump (SLJ) test for measuring leaping distance; the plate tapping (PTT) for evaluating movement speed; the obstacle course backwards (OCB) for assessing body coordination; and the shuttle run test 4 × 5 m (SRT) for measuring speed and agility.

INTERVENTIONS:
Other: Traditional Play — The intervention for the traditional play group included activities such as Shtapu and skipping rope. Both traditional play activities were scheduled 3 times per week (3 Session/week) over the 6-month period.
  Both activities took place outdoors and in the institutional gymnasium, depending on the prevailing weather conditions. Each session lasted 35 minutes and took place in the morning hours (8-11 a.m.). Prior to each type of activity, a specific warm-up was conducted, following methodological guidelines for preschoolers' physical education.
  Arms: Traditional Play

SUMMARY:
Childhood play is crucial for the comprehensive development of children, as it fosters social and emotional skills. This study examines the relative effects of conventional games versus unstructured play on the social interaction and physical fitness of elementary school students. This study aims to explore the impact of traditional games and free play on motor fitness and social interaction among primary school children and also seeks to offer insights into how these activities can benefit physical health and social development in the school environment. A randomized clinical trial will be conducted to evaluate the comparative effects of traditional play and free play on motor fitness and social interaction in primary school children. Study will include 104 children with aged 5 to 9 and take place in Sukkur schools for a duration of 10 months.

Traditional play groups and free play groups. The Social Skills Rating Scale (SSRS) will be utilized to evaluate social interaction. The statistical software SPSS version 27.00 will be used to analyze the data.

DETAILED DESCRIPTION:
Childhood play is crucial for the comprehensive development of children, as it fosters social and emotional skills that equip them to face challenges throughout their lives, from infancy to adulthood. This study examines the relative effects of conventional games versus unstructured play on the social interaction and physical fitness of elementary school students. Traditional games, marked by organized rules, and free play, characterized by spontaneous, unstructured activities, are represented by different types of play that affect social behaviors and motor skills.

Understanding these effects is essential, as participating in physical activities not only boosts physical health but also influences cognitive and social skills, which are important for long-term mental and physical well-being. This study aims to explore the impact of traditional games and free play on motor fitness and social interaction among primary school children and also seeks to offer insights into how these activities can benefit physical health and social development in the school environment. A randomized clinical trial will be conducted to evaluate the comparative effects of traditional play and free play on motor fitness and social interaction in primary school children. This study will include children aged 5 to 9 and take place in Sukkur schools for a duration of 10 months.

Traditional play groups will partake in organized conventional activities that are included in their schedule, while free play groups will involve themselves in unregulated spontaneous play. The participants will be segregated into 2 distinct groups. The flamingo balance tests (FLA) will be used to assess motor fitness related to balance; the standing long jump (SLJ) test for measuring leaping distance; the plate tapping (PTT) for evaluating movement speed; the obstacle course backwards (OCB) for assessing body coordination; and the shuttle run test 4 × 5 m (SRT) for measuring speed and agility. The Social Skills Rating Scale (SSRS) will be utilized to evaluate social interaction. The statistical software SPSS version 27.00 will be used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be within the age range of 5 to 9 years.
* Currently enrolled in a primary school program.
* Both male and female participants are included.
* Participants must have parental or guardian consent to participate in the study.
* Participants must be regularly attending primary school without prolonged absences

Exclusion Criteria:

* Musculoskeletal disorders (e.g., poliomyelitis, muscular dystrophy).
* Neurological disorders (e.g., epilepsy, developmental delay).
* Orthopedic disorders (e.g., fractures, joint disorders).
* Diabetes or other metabolic syndrome conditions.
* Chronic health conditions affecting physical activity participation.
* Engaged in organized sports or structured physical activities outside of the primary school curriculum

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Social Skills Rating Scale (SSRS) | 6 week
  Surveys measuring social skills from kindergarten through the 12th grade are conducted through the Social Skills Rating System. In the SSRS there are 3 rating forms are included: teacher, parent, and student. Problem behavior is evaluated by the teacher and parent forms, with a special emphasis on externalizing problems, internalizing problems, and hyperactivity issues. Lastly, the teacher form assesses motivation, parental support, reading and math proficiency, as well as cognitive functioning in order to determine academic competency

CONTACTS AND LOCATIONS:
Overall Officials: Maria Amjad, MSPT(Peads), Principal Investigator — Riphah International University
Locations (1):
- School of Sindh, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No